CLINICAL TRIAL: NCT00045422
Title: A Phase II Open Label Study to Determine Safety and Efficacy of Interferon-alpha in Combination With Imantinib Mesylate (Gleevec) in Patients With Chronic Phase Chronic Myelogenous Leukemia Who Have Not Achieved a Complete Cytogenetic Response to Gleevec as a Single Agent
Brief Title: Interferon Alfa and Imatinib Mesylate in Treating Patients With Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 02-013; CDR0000256469 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2105
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia, BCR-ABL1 positive; chronic phase chronic myelogenous leukemia; childhood chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Interferon-alpha; Imatinib Mesylate

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Combining interferon alfa with imatinib mesylate may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining interferon alfa with imatinib mesylate in treating patients who have chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether interferon alfa in combination with imatinib mesylate adds to the hematologic, cytogenetic, and molecular response rates in patients with chronic phase chronic myelogenous leukemia that is newly diagnosed or has not achieved a complete cytogenetic response to imatinib mesylate alone.

OUTLINE: Patients receive oral imatinib mesylate (STI-571) once daily for 9 months. At 9 months, patients with more than 35% Philadelphia chromosome-positive (Ph+) cells in bone marrow receive oral STI-571 twice daily for 3 more months. At 12 months, patients with more than 35% Ph+ cells in bone marrow receive oral STI-571 once daily and interferon alfa subcutaneously once daily. Treatment continues for at least 1 year in the absence of disease progression or unacceptable toxicity. Patients with an appropriate HLA-matched donor may choose to have a bone marrow transplantation at any time during the study.

Patients are followed every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 80 patients (60 without an HLA-matched donor and 20 with an HLA-matched donor) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of chronic phase chronic myelogenous leukemia

  * Cytogenetically confirmed Philadelphia chromosome-positive disease or other variant of t(9;22)

    * No secondary chromosomal abnormalities
  * No more than 10% blasts in bone marrow
  * Newly diagnosed OR
  * Received prior imatinib mesylate as a single agent for no more than the past 9 months without achieving a complete cytogenetic response
* No evidence of extramedullary involvement except nodes, liver, or spleen

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-3

Life expectancy

* Not specified

Hematopoietic

* Platelet count greater than 100,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT no greater than 2 times ULN
* INR no greater than 1.5 times ULN*
* PTT no greater than 1.5 times ULN* NOTE: * Except patients on anticoagulants

Renal

* Creatinine no greater than 2 times ULN

Other

* Considered potentially reliable
* No history of noncompliance to medical regimens
* No other active malignancy requiring chemotherapy or radiotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior interferon therapy
* No prior stem cell or bone marrow transplantation

Chemotherapy

* No prior chemotherapy (except hydroxyurea and/or anagrelide to control counts)

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* At least 4 weeks since prior major surgery and recovered

Other

* No concurrent grapefruit juice or grapefruit products
* No concurrent warfarin
* Concurrent low-molecular weight heparin allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellin Berman, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States